CLINICAL TRIAL: NCT00861705
Title: Randomized Phase II 2 x 2 Factorial Trial of the Addition of Carboplatin +/- Bevacizumab to Neoadjuvant Weekly Paclitaxel Followed by Dose-Dense AC in Hormone Receptor-Poor/HER2-Negative Resectable Breast Cancer
Brief Title: Paclitaxel With or Without Carboplatin and/or Bevacizumab Followed by Doxorubicin and Cyclophosphamide in Treating Patients With Breast Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01172; NCI-2009-01172 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CALGB 40603/CTSU 40603; CALGB-40603; CDR0000636850; CALGB 40603 (Other: Alliance for Clinical Trials in Oncology); CALGB-40603 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Male Breast Carcinoma; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage IIIA Breast Cancer AJCC v7; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Carboplatin; Cyclophosphamide; Doxorubicin; Paclitaxel; Taxes

ARMS (4):
- Arm I (paclitaxel, doxorubicin, cyclophosphamide) (Active Comparator): Patients receive paclitaxel IV over 60 minutes once weekly in weeks 1-12. Patients then receive dose-dense doxorubicin hydrochloride IV over 5-10 minutes and cyclophosphamide IV over 5-30 minutes (ddAC) once in weeks 13, 15, 17, and 19.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel
- Arm II (paclitaxel, ddAC, bevacizumab) (Experimental): Patients receive paclitaxel and ddAC as in Arm I. Patients also receive bevacizumab IV over 30-90 minutes in weeks 1, 3, 5, 7, 9, 11, 13, 15, and 17.
  Interventions: Biological: Bevacizumab; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel
- Arm III (paclitaxel, ddAC, carboplatin) (Experimental): Patients receive paclitaxel and ddAC as in Arm I. Patients also receive carboplatin IV over 30 minutes once in weeks 1, 4, 7, and 10.
  Interventions: Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel
- Arm IV (paclitaxel, ddAC, bevacizumab, carboplatin) (Experimental): Patients receive paclitaxel and ddAC as in Arm I, bevacizumab as in Arm II, and carboplatin as in Arm III.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm II (paclitaxel, ddAC, bevacizumab); Arm IV (paclitaxel, ddAC, bevacizumab, carboplatin)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm III (paclitaxel, ddAC, carboplatin); Arm IV (paclitaxel, ddAC, bevacizumab, carboplatin)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This randomized phase II trial studies how well paclitaxel with or without carboplatin and/or bevacizumab followed by doxorubicin and cyclophosphamide works in treating patients with breast cancer that can be removed by surgery. Drugs used in chemotherapy, such as paclitaxel, carboplatin, doxorubicin, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Bevacizumab may stop the growth of tumor cells by blocking blood flow to the tumor. Giving chemotherapy together with bevacizumab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether adding bevacizumab to neoadjuvant weekly paclitaxel (+/- carboplatin) and subsequent dose-dense doxorubicin and cyclophosphamide (ddAC) significantly raises the rate of pathologic complete response (pCR) in the breast in patients with hormone receptor (HR)-poor/human epidermal growth factor receptor 2 (HER2) (-), resectable breast cancer.

II. To determine whether adding carboplatin every 3 weeks to neoadjuvant weekly paclitaxel followed by ddAC (+/- bevacizumab) significantly raises the rate of pCR in the breast in patients with HR-poor/HER2(-), resectable breast cancer.

III. To determine whether adding bevacizumab every 2 weeks to neoadjuvant weekly paclitaxel (+/- carboplatin) and subsequent ddAC significantly raises the rate of pCR in the breast in patients with basal-like breast cancers, as defined by gene expression array.

IV. To determine whether adding carboplatin every 3 weeks to neoadjuvant weekly paclitaxel followed by ddAC (+/- bevacizumab) significantly raises the rate of pCR in the breast in patients with basal-like breast cancers, as defined by gene expression array.

SECONDARY OBJECTIVES:

I. To determine the pCR rates in the breast and axilla, using American Joint Committee On Cancer (AJCC) TNM criteria (version 6), to neoadjuvant weekly paclitaxel, with or without carboplatin, followed by ddAC, with or without bevacizumab, given concurrently with the weekly paclitaxel and ddAC, in (a) patients with HR-poor/HER2(-), resectable breast cancer and (b) the subset of patients with basal-like breast cancers, as defined by gene expression array.

II. To assess whether there is an interaction between the addition of carboplatin and bevacizumab to neoadjuvant chemotherapy (NAC) with weekly paclitaxel followed by ddAC as regards the path pCR rates in (a) patients with HR-poor/HER2(-), resectable breast cancer and (b) the subset of patients with basal-like breast cancers, as defined by gene expression array.

III. To assess the toxicity of the control regimen (weekly paclitaxel followed by ddAC) and any incremental toxicities associated with the addition of carboplatin and/or bevacizumab in this patient population, including the incidence of febrile neutropenia, grade >= 3 thrombocytopenia, grade >= 2 neurotoxicity, grade >= 3 hypertension, and clinically significant bleeding or thrombotic (including cardiovascular and cerebrovascular) events.

IV. To determine the recurrence-free survival (RFS) measured from definitive surgery to first event, and time to first failure (TFF) measured from study entry to first event.

V. To determine overall survival (OS), defined as time from registration to death from any cause.

VI. To assess the impact of NAC with weekly paclitaxel followed by ddAC, with or without carboplatin and/or bevacizumab, on axillary lymph node involvement at surgery, particularly in patients with clinically or histologically positive axillary lymph nodes prior to initiation of NAC.

VII. To assess the impact of the addition of bevacizumab to NAC on the incidence and severity of post-op complications, especially excessive bleeding, delayed wound healing, and thrombotic complications.

VIII. To evaluate residual cancer burden (RCB) as a predictor of RFS, TFF and OS.

IX. To determine the correlation between clinical, radiographic, and pathologic response.

TERTIARY OBJECTIVES:

I. To assess whether the impact of the addition of carboplatin and/or bevacizumab to NAC with weekly paclitaxel followed by ddAC on achievement of pathologic CRs in patients with HR-poor/HER2(-), resectable breast cancer is influenced by molecular subtype, as defined by gene expression array.

II. To obtain blood, fresh frozen and fixed tumor tissue to test specific hypotheses for which biomarker data exist and to evaluate biomarkers in tissue, blood, and serum that may influence response to and toxicity of weekly paclitaxel, ddAC, carboplatin, and/or bevacizumab.

III. To obtain blood samples to test specific hypotheses for which biomarker data exist and to evaluate biomarkers in blood that may influence response to and toxicity of weekly paclitaxel, ddAC, carboplatin and/or bevacizumab.

IV. To determine the surgical practice patterns for breast conservation and sentinel lymphadenectomy in patients undergoing neoadjuvant chemotherapy.

V. To examine the practice patterns and use of sentinel lymphadenectomy (pre-chemotherapy or post-chemotherapy) in patients with T2 or T3 breast cancer.

VI. To examine the proportion of patients who presented with T2 or T3 cancers who undergo mastectomy despite cytoreduction adequate for breast conservation.

VII. To determine the radiotherapy practice patterns for post-mastectomy and regional nodal irradiation in patients undergoing neoadjuvant chemotherapy.

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 60 minutes once weekly in weeks 1-12. Patients then receive dose-dense doxorubicin hydrochloride IV over 3-10 minutes and cyclophosphamide IV over 5-60 minutes (ddAC) once in weeks 13, 15, 17, and 19.

ARM II: Patients receive paclitaxel and ddAC as in Arm I. Patients also receive bevacizumab IV over 30-90 minutes once in weeks 1, 3, 5, 7, 9, 11, 13, 15, and 17.

ARM III: Patients receive paclitaxel and ddAC as in Arm I. Patients also receive carboplatin IV over 30 minutes once in weeks 1, 4, 7, and 10.

ARM IV: Patients receive paclitaxel and ddAC as in Arm I, bevacizumab as in Arm II, and carboplatin as in Arm III.

Patients in all arms undergo definitive surgery (i.e., modified radical mastectomy or breast-conserving surgery with appropriate management of the axilla) between 4-8 weeks after completion of neoadjuvant therapy.

After completion of study treatment, patients are followed up periodically for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer, diagnosed by core needle or incisional biopsy (excisional biopsy not permitted)
* The invasive tumor must be hormone receptor-poor, defined as both estrogen receptor (ER) and progesterone receptor (PgR) negative or staining present in =< 10% of invasive cancer cells by immunohistochemistry (IHC)
* The invasive tumor must be HER2-negative, defined as IHC 0-1+ or with a fluorescent in situ hybridization (FISH) ratio (HER2 gene copy/chromosome 17) of < 2.0 if IHC 2+
* Clinical stage II-III invasive breast cancer with intent to perform surgical resection after neoadjuvant therapy; patients with inflammatory breast cancer are not eligible; staging to rule out metastatic disease is recommended for clinical stage III patients
* Patients with multicentric or bilateral disease are eligible if the target lesion meets eligibility criteria
* Patient agrees to undergo pretreatment research biopsies
* No prior chemotherapy, hormone therapy, or radiation therapy with therapeutic intent for this cancer
* The target lesion in the breast must be >= 1 cm, clinically or radiographically; palpable or radiographically measurable axillary adenopathy will be recorded but will not serve as measurable disease for the primary endpoint; patients with axillary disease only (no identifiable tumor in the breast that is >= 1 cm on physical exam or radiographic study) are not eligible to participate
* Patients with a history of significant bleeding episodes (e.g., hemoptysis, upper or lower gastrointestinal [GI] bleeding) within 6 months of registration are not eligible
* No serious or non-healing wound, skin ulcers or bone fracture; no abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within the past 6 months; no major surgical procedure within 28 days prior to randomization or anticipation of need for major surgery during the course of study
* The following are not considered to be major surgical procedures that would be prohibited in the 28 days prior to, or following study randomization: obtaining the required research needle biopsies; placement of a radiopaque clip to localize a tumor or tumors for subsequent surgical resection; placement of a port for central venous access; fine needle aspiration of a prominent or suspicious axillary lymph node; needle biopsy of a clinically or radiographically detected lesion to rule out metastatic disease; or pretreatment sentinel lymph node sampling
* No baseline neuropathy grade >= 2
* Zubrod performance status 0-1
* Pregnant or nursing women are not eligible; all women of reproductive potential must have a negative pregnancy test at baseline and agree to use an effective, non-hormonal method of contraception during the entire period of treatment on the study
* Patients with congestive heart failure are not eligible, nor are patients with myocardial infarction, unstable angina pectoris, an arterial thrombotic event, stroke or transient ischemia attack (TIA) within the past 12 months, uncontrolled hypertension (systolic blood pressure [SBP] > 160 or diastolic blood pressure [DBP] > 90), uncontrolled or symptomatic arrhythmia, or grade II or greater peripheral vascular disease
* Patients must have a pretreatment multi gated acquisition (MUGA) scan or echocardiogram with a left ventricular ejection fraction (LVEF) above the institutional lower limit of normal
* Granulocytes > 1,000/mcl
* Platelets > 100,000/mcl
* Total bilirubin =< 1.5 x upper limits of normal
* Calculated or measured > 30 ml/min
* Urine protein =< 1+ or urine protein to creatinine (UPC) ratio < 1

  * Patients discovered to have >= 2+ proteinuria at baseline must undergo a 24-hour urine collection that must demonstrate < 1 g of protein/24 hr, or UPC ratio < 1 to allow participation in the study
* Serum alanine aminotransferase (ALT) =< 2.5 x upper limits of normal
* Serum beta human chorionic gonadotropin (HCG) negative (for women of child bearing potential)
* Prothrombin time (PT)/international normalized ratio (INR) =< 1.5 x upper limit of normal (ULN)

  * Unless patient is on therapeutic doses of warfarin; if so, the patient must have an INR =< 3 on a stable dose of warfarin, must have not active bleeding or pathologic condition that is associated with a high risk of bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2009-07-21 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2025-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William M Sikov, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (448):
- United States (448):
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Wilma Chan Highland Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Salinas Valley Memorial, Salinas, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Breastlink Medical Group Inc, Santa Ana, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Cancer Center of South Florida-Lake Worth, Lake Worth, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - HaysMed, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - AdventHealth Shawnee Mission, Shawnee Mission, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Eastern Maine Medical Center, Bangor, Maine
  - New England Cancer Specialists, Westbrook, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - Coney Island Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Queens Hospital Center, Jamaica, New York
  - Garnet Health Medical Center, Middletown, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Nash UNC HealthCare, Rocky Mount, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Saint Mary's Medical Center, Huntington, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Fox Valley Surgical Associates Limited, Appleton, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Cancer Care-Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Glendale, Glendale, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.

REFERENCES:
- [Derived] Shepherd JH, Ballman K, Polley MC, Campbell JD, Fan C, Selitsky S, Fernandez-Martinez A, Parker JS, Hoadley KA, Hu Z, Li Y, Soloway MG, Spears PA, Singh B, Tolaney SM, Somlo G, Port ER, Ma C, Kuzma C, Mamounas E, Golshan M, Bellon JR, Collyar D, Hahn OM, Hudis CA, Winer EP, Partridge A, Hyslop T, Carey LA, Perou CM, Sikov WM. CALGB 40603 (Alliance): Long-Term Outcomes and Genomic Correlates of Response and Survival After Neoadjuvant Chemotherapy With or Without Carboplatin and Bevacizumab in Triple-Negative Breast Cancer. J Clin Oncol. 2022 Apr 20;40(12):1323-1334. doi: 10.1200/JCO.21.01506. Epub 2022 Jan 19. PMID 35044810
- [Derived] Sikov WM, Berry DA, Perou CM, Singh B, Cirrincione CT, Tolaney SM, Kuzma CS, Pluard TJ, Somlo G, Port ER, Golshan M, Bellon JR, Collyar D, Hahn OM, Carey LA, Hudis CA, Winer EP. Impact of the addition of carboplatin and/or bevacizumab to neoadjuvant once-per-week paclitaxel followed by dose-dense doxorubicin and cyclophosphamide on pathologic complete response rates in stage II to III triple-negative breast cancer: CALGB 40603 (Alliance). J Clin Oncol. 2015 Jan 1;33(1):13-21. doi: 10.1200/JCO.2014.57.0572. Epub 2014 Aug 4. PMID 25092775
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 (Pac --> ddAC): Patients receive paclitaxel (pac) IV over 60 minutes once weekly in weeks 1-12. Patients then receive dose-dense doxorubicin hydrochloride IV over 5-10 minutes and cyclophosphamide IV over 5-30 minutes (ddAC) once in weeks 13, 15, 17, and 19.
  doxorubicin hydrochloride: Given IV
  paclitaxel: Given IV
  cyclophosphamide: Given IV
- Arm 2 (Pac + Bev --> ddAC + Bev): Patients receive pac and ddAC as in arm 1. Patients also receive bevacizumab (bev) IV over 30-90 minutes in weeks 1, 3, 5, 7, 9, 11, 13, 15, and 17.
  doxorubicin hydrochloride: Given IV
  paclitaxel: Given IV
  cyclophosphamide: Given IV
  bevacizumab: Given IV
- Arm 3 (Pac + Carboplatin --> ddAC): Patients receive pac and ddAC as in arm 1. Patients also receive carboplatin IV over 30 minutes once in weeks 1, 4, 7, and 10.
  doxorubicin hydrochloride: Given IV
  paclitaxel: Given IV
  cyclophosphamide: Given IV
  carboplatin: Given IV
- Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev): Patients receive pac and ddAC as in arm 1, bev as in arm 2, and carboplatin as in arm 3.
  doxorubicin hydrochloride: Given IV
  paclitaxel: Given IV
  cyclophosphamide: Given IV
  bevacizumab: Given IV
  carboplatin: Given IV
Period: Overall Study
Arm/Group | Arm 1 (Pac --> ddAC) | Arm 2 (Pac + Bev --> ddAC + Bev) | Arm 3 (Pac + Carboplatin --> ddAC) | Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev)
Started | 115 | 113 | 113 | 113
Completed | 108 | 110 | 113 | 112
Not Completed | 7 | 3 | 0 | 1
Not completed — Never Began Treatment | 7 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Using a modified intent-to-treat approach only patients who began protocol treatment (n=443) were included in analyses for neoadjuvant treatment and toxicity. Analyses for surgical endpoints excluded 10 patients who withdrew consent prior to surgery (n=433). All analyses considered patients according to treatment assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Pac --> ddAC) | Arm 2 (Pac + Bev --> ddAC + Bev) | Arm 3 (Pac + Carboplatin --> ddAC) | Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev) | Total
Number analyzed (Participants) | 115 | 113 | 113 | 113 | 454
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (11.1) | 48.3 (10.8) | 50.9 (10.8) | 47.1 (9.8) | 49.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 113 | 113 | 113 | 454
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 2 | 3
  Asian | 1 | 5 | 4 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 20 | 21 | 27 | 21 | 89
  White | 86 | 84 | 80 | 81 | 331
  More than one race | 1 | 1 | 1 | 2 | 5
  Unknown or Not Reported | 5 | 2 | 1 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) in the Breast. Defined as the Absence of Residual Invasive Carcinoma in the Breast (ypT0/is).
Description: Assessment of the difference in percentage of participants with pCR in the breast between regimens that contain carboplatin (arms 3&4) versus not (arms 1&2) will use a one-sided chi square test. 95% confidence intervals around the incidence of pCR will also be constructed using exact binomial methods.
Time Frame: At the time of definitive surgical removal, up to 28 weeks
Population: All patients who began protocol neoadjuvant therapy and are assessable for pCR endpoint (N=433).
Measure: Number (95% Confidence Interval); unit: percentage of participants with pCR
Groups:
- Factor A: Carboplatin: Factor A is the addition or not of carboplatin: the experimental regimens included carboplatin (Arms 3 & 4).
- Factor A: No Carboplatin: Factor A is the addition or not of carboplatin; the control regimens did not include carboplatin (Arms 1 & 2).
Arm/Group | Factor A: Carboplatin | Factor A: No Carboplatin
Number analyzed (Participants) | 221 | 212
percentage of participants with pCR | 60 [54 to 66] | 46 [40 to 53]
Statistical Analysis 1: Comparison: Factor A: Carboplatin vs Factor A: No Carboplatin; The study was designed to detect an increase in the incidence of pCR from 35% in the control arm to 55% in the experimental arm using a 1-sided chi square test of proportions. With a target sample of 362 patients and assuming a 10% dropout rate, an overall assessable sample size of 326 patients resulted in > 95% power; Test type: Superiority or Other; p = 0.0018, Chi-squared; Reported p-values are unadjusted and 1-sided

2. Primary Outcome: Pathologic Complete Response (pCR) in the Breast. Defined as the Absence of Residual Invasive Carcinoma in the Breast (ypT0/is).
Description: Assessment of the difference in percentage of participants with pCR in the breast between regimens that contain bevacizumab (arms 2&4) versus not (arms 1&3) will use a one-sided chi square test. 95% confidence intervals around the incidence of pCR will also be constructed using exact binomial methods.
Time Frame: At the time of definitive surgical removal, up to 28 weeks
Population: All patients who began protocol neoadjuvant therapy and are assessable for pCR endpoint (N=433).
Measure: Number (95% Confidence Interval); unit: percentage of participants with pCR
Groups:
- Factor B: Bevacizumab: Factor B is the addition or not of bevacizumab: the experimental regimens included bevacizumab (Arms 2 & 4).
- Factor B: No Bevacizumab: Factor B is the addition or not of bevacizumab: the control regimens did not include bevacizumab (Arms 1 & 3)
Arm/Group | Factor B: Bevacizumab | Factor B: No Bevacizumab
Number analyzed (Participants) | 215 | 218
percentage of participants with pCR | 59 [52 to 65] | 48 [41 to 54]
Statistical Analysis 1: Comparison: Factor B: Bevacizumab vs Factor B: No Bevacizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0089, Chi-squared; Reported p-values are unadjusted and 1-sided

3. Secondary Outcome: Pathologic Complete Response (pCR) in the Breast and Axilla. Defined as the Absence of Residual Invasive Carcinoma in the Breast (ypT0/is) Plus the Absence of Any Tumor Deposit >0.2 mm in Sampled Axillary Nodes (ypT0/isN0).
Description: Comparing regimens that contain carboplatin (arms 3&4) versus not (arms 1&2).
Time Frame: At the time of definitive surgical removal, up to 28 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants with pCR
Arm/Group | Factor A: Carboplatin | Factor A: No Carboplatin
Number analyzed (Participants) | 221 | 212
percentage of participants with pCR | 54 [48 to 61] | 41 [35 to 48]
Statistical Analysis 1: Comparison: Factor A: Carboplatin vs Factor A: No Carboplatin; Test type: Superiority or Other; p = 0.0029, Chi-squared; Reported p-values are unadjusted and 1-sided

4. Secondary Outcome: Pathologic Complete Response (pCR) in the Breast and Axilla. Defined as the Absence of Residual Invasive Carcinoma in the Breast (ypT0/is) Plus the Absence of Any Tumor Deposit >0.2 mm in Sampled Axillary Nodes (ypT0/isN0).
Description: Comparing regimens that contain bevacizumab (arms 2&4) versus not (arms 1&3).
Time Frame: At the time of definitive surgical removal, up to 28 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants with pCR
Arm/Group | Factor B: Bevacizumab | Factor B: No Bevacizumab
Number analyzed (Participants) | 215 | 218
percentage of participants with pCR | 52 [45 to 58] | 44 [38 to 51]
Statistical Analysis 1: Comparison: Factor B: Bevacizumab vs Factor B: No Bevacizumab; Test type: Superiority or Other; p = 0.057, Chi-squared; Reported p-values are unadjusted and 1-sided

5. Secondary Outcome: Pathologic Stage in the Breast and in the Breast Plus Axilla as Measured by American Joint Committee on Cancer (AJCC) Tumor Node Metastasis (TNM) Staging Criteria (Version 6)
Description: Stage II is (T2,T3, N0, M0) tumor size more than 2 cm but no deep extradermal structure invasion, no regional lymph node metastasis, and no distant metastasis. Stage III is (T4, N0, M0) tumor invasion of deep extradermal structures, no regional lymph node metasis, and no distant metasasis or (Any T, N1, M0) Any tumor size, regional lymph node metastasis, and no distant metastasis.
Time Frame: at definitive surgery, up to 28 weeks
Measure: Number; unit: participants
Arm/Group | Arm 1 (Pac --> ddAC) | Arm 2 (Pac + Bev --> ddAC + Bev) | Arm 3 (Pac + Carboplatin --> ddAC) | Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev)
Number analyzed (Participants) | 107 | 105 | 111 | 110
participants
  Breast : Stage II | 42 | 49 | 51 | 70
  Breast : Stage III | 42 | 55 | 57 | 62
  Breast/Axilla : Stage II | 41 | 42 | 47 | 63
  Breast/Axilla : Stage III | 36 | 45 | 51 | 54

6. Secondary Outcome: Radiographic Response Assessed by Tumor Measurement
Description: Assessed by RECIST, each patient will have a pre-therapy baseline radiographic tumor measurement, preferably by MRI, however if logistic or practical or financial issues preclude MRI use, mammogram or ultrasound may be substituted. The longest diameter (LD) of the target lesion at the time of study initiation will be reported as the baseline LD. The baseline LD of the target lesion will be used as reference to further characterize the objective tumor response of the measurable dimension of the disease. Radiographic complete response: Disappearance of the target lesion. Radiographic partial response (PR): At least a 30% decrease in the longest diameter (LD) of the target lesion taking as reference the baseline LD.
Time Frame: Baseline; at completion of neoadjuvant therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Pac --> ddAC) | Arm 2 (Pac + Bev --> ddAC + Bev) | Arm 3 (Pac + Carboplatin --> ddAC) | Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev)
Number analyzed (Participants) | 108 | 110 | 112 | 112
Participants
  Complete Response | 11 | 12 | 19 | 13
  Partial Response | 16 | 11 | 16 | 17
  Failures | 81 | 87 | 77 | 82

7. Secondary Outcome: Clinical Response Assessed by Tumor Measurement
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST). Both target and, in the event of multifocal or multicentric invasive breast cancer, nontarget lesions should be followed clinically and their clinical size recorded at aseline. Measurements thereafter are required at the completion of 12 weeks of paclitaxel or paclitaxel/carboplatin and at the completion of all neoadjuvant chemotherapy. At any time point, these lesions should be categorized regarding whether there is evidence of progression. If "yes", the study chair should be notified in order to determine whether the patient should come off protocol treatment. In-situcarcinoma does not represent a non-target lesion and should not be recorded or followed.
Time Frame: Baseline; at completion of neoadjuvant therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Pac --> ddAC) | Arm 2 (Pac + Bev --> ddAC + Bev) | Arm 3 (Pac + Carboplatin --> ddAC) | Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev)
Number analyzed (Participants) | 108 | 110 | 112 | 112
Participants
  Complete Response | 28 | 35 | 45 | 40
  Partial Response | 37 | 38 | 36 | 37
  Failures | 43 | 37 | 31 | 35

8. Secondary Outcome: Overall Survival
Description: Number of Participants who Died Due to Any Cause
Time Frame: up to 10 years
Population: All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Pac --> ddAC) | Arm 2 (Pac + Bev --> ddAC + Bev) | Arm 3 (Pac + Carboplatin --> ddAC) | Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev)
Number analyzed (Participants) | 107 | 110 | 112 | 112
Participants | 22 | 26 | 30 | 24
Statistical Analysis 1: Comparison: Arm 1 (Pac --> ddAC) vs Arm 2 (Pac + Bev --> ddAC + Bev); Test type: Superiority; Cox Proportional Hazard = 1.19, 95% CI 2-sided [0.67 to 2.10]
Statistical Analysis 2: Comparison: Arm 1 (Pac --> ddAC) vs Arm 3 (Pac + Carboplatin --> ddAC); Test type: Superiority; Cox Proportional Hazard = 1.43, 95% CI 2-sided [0.82 to 2.47]
Statistical Analysis 3: Comparison: Arm 1 (Pac --> ddAC) vs Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev); Test type: Superiority; Cox Proportional Hazard = 0.82, 95% CI 2-sided [0.49 to 1.37]

9. Secondary Outcome: Recurrence-free Survival
Description: From definitive surgery to first instance of ipsilateral invasive breast tumor recurrence, local/regional invasive breast cancer recurrence, distant recurrence, or death from any cause. Number of Participants who Died Due to Any Cause or had a recurrence.
Time Frame: up to 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Pac --> ddAC) | Arm 2 (Pac + Bev --> ddAC + Bev) | Arm 3 (Pac + Carboplatin --> ddAC) | Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev)
Number analyzed (Participants) | 108 | 110 | 112 | 112
Participants
  With event | 32 | 34 | 37 | 27
  Without event | 76 | 76 | 75 | 85
Statistical Analysis 1: Comparison: Arm 1 (Pac --> ddAC) vs Arm 2 (Pac + Bev --> ddAC + Bev); Test type: Superiority; Cox Proportional Hazard = 1.08, 95% CI 2-sided [0.66 to 1.75]
Statistical Analysis 2: Comparison: Arm 1 (Pac --> ddAC) vs Arm 3 (Pac + Carboplatin --> ddAC); Test type: Superiority; Cox Proportional Hazard = 1.20, 95% CI 2-sided [0.74 to 1.92]
Statistical Analysis 3: Comparison: Arm 1 (Pac --> ddAC) vs Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev); Test type: Superiority; Cox Proportional Hazard = 0.82, 95% CI 2-sided [0.49 to 1.37]

10. Secondary Outcome: Count of Participants With a First Failure, Defined as First Instance of Ipsilateral Invasive Breast Tumor Recurrence, Local/Regional Invasive Breast Cancer Recurrence, Distant Recurrence, or Death From Any Cause
Description: From study entry to first event.
Time Frame: up to 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Pac --> ddAC) | Arm 2 (Pac + Bev --> ddAC + Bev) | Arm 3 (Pac + Carboplatin --> ddAC) | Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev)
Number analyzed (Participants) | 108 | 110 | 112 | 112
Participants
  With event | 23 | 26 | 28 | 22
  Without event | 85 | 84 | 84 | 90
Statistical Analysis 1: Comparison: Arm 1 (Pac --> ddAC) vs Arm 2 (Pac + Bev --> ddAC + Bev); Test type: Superiority; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.66 to 2.03]
Statistical Analysis 2: Comparison: Arm 1 (Pac --> ddAC) vs Arm 3 (Pac + Carboplatin --> ddAC); Test type: Superiority; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.72 to 2.16]
Statistical Analysis 3: Comparison: Arm 1 (Pac --> ddAC) vs Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev); Test type: Superiority; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.53 to 1.70]

11. Secondary Outcome: Incidence and Severity of Post-op Complications, Namely Excessive Bleeding, Delayed Wound Healing, and Wound Dehiscence.
Description: Assessed by physician observation.
Time Frame: at definitive surgery, up to 28 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants with event
Arm/Group | Factor B: Bevacizumab | Factor B: No Bevacizumab
Number analyzed (Participants) | 213 | 214
percentage of participants with event
  Excessive bleeding | 0 [0 to 2] | 0 [0 to 3]
  Delayed healing | 1 [0 to 3] | 0 [0 to 3]
  Wound dehiscence | 1 [1 to 4] | 0 [0 to 3]

ADVERSE EVENTS:
Description: Out of the 454 participants, 443 began treatment. Six participants were not evaluable for adverse events due to site non-compliance (2 in Arm 2 and 4 in Arm 3). Therefore, adverse events data are available for 437 participants (108 in Arm 1, 108 in Arm 2, 109 in Arm 3, and 112 in Arm 4).
Groups:
- Arm 1 (Pac --> ddAC): cyclophosphamide: Given IV
- Arm 2 (Pac + Bev --> ddAC + Bev): bevacizumab: Given IV
- Arm 3 (Pac + Carboplatin --> ddAC); Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev): carboplatin: Given IV
Arm/Group | Arm 1 (Pac --> ddAC) | Arm 2 (Pac + Bev --> ddAC + Bev) | Arm 3 (Pac + Carboplatin --> ddAC) | Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev)
Serious Adverse Events (participants affected / at risk) | 15/108 | 27/108 | 21/109 | 39/112
Other Adverse Events (participants affected / at risk) | 107/108 | 104/108 | 106/109 | 109/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Pac --> ddAC) (N=108) | Arm 2 (Pac + Bev --> ddAC + Bev) (N=108) | Arm 3 (Pac + Carboplatin --> ddAC) (N=109) | Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev) (N=112)
Blood disorder (Blood and lymphatic system disorders) | 11 (11) | 14 (17) | 17 (20) | 28 (33)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 4 (5) | 9 (9) | 15 (16)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 4 (5) | 6 (6)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 6 (7)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 9 (11) | 3 (4) | 18 (19)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 6 (6) | 7 (7) | 14 (15)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 5 (6) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 8 (9)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Ileal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 5 (5) | 4 (5) | 8 (8)
Nausea (Gastrointestinal disorders) | 6 (6) | 13 (15) | 11 (12) | 21 (23)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 7 (7) | 5 (6) | 15 (16)
Chest pain (General disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Chills (General disorders) | 1 (1) | 2 (2) | 3 (3) | 3 (4)
Edema limbs (General disorders) | 3 (3) | 3 (4) | 2 (2) | 2 (3)
Fatigue (General disorders) | 12 (12) | 22 (25) | 19 (22) | 36 (41)
Fever (General disorders) | 3 (3) | 3 (3) | 5 (5) | 3 (3)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General symptom (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 4 (5) | 4 (5) | 5 (5)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Catheter related infection (Infections and infestations) | 1 (1) | 5 (5) | 1 (2) | 2 (2)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 1 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 5 (5)
Uterine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 4 (4) | 4 (5) | 9 (9)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 3 (3) | 6 (6)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 4 (5) | 8 (8)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cardiac troponin T increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Haptoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Leukocyte count decreased (Investigations) | 6 (6) | 6 (7) | 13 (15) | 14 (15)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 1 (1) | 5 (6) | 7 (7)
Neutrophil count decreased (Investigations) | 7 (7) | 12 (15) | 16 (18) | 22 (26)
Platelet count decreased (Investigations) | 6 (6) | 8 (10) | 16 (18) | 21 (25)
Weight loss (Investigations) | 1 (1) | 5 (5) | 2 (2) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 6 (7) | 8 (10) | 11 (12)
Blood glucose increased (Metabolism and nutrition disorders) | 5 (5) | 5 (6) | 7 (8) | 10 (11)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 4 (4) | 8 (8)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 4 (4) | 9 (10)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (4) | 5 (6) | 5 (5) | 8 (9)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (6) | 7 (7)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (3) | 6 (6) | 7 (7) | 7 (8)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 5 (5) | 10 (11)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abdominal soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (3) | 2 (3)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 1 (1) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5) | 3 (3) | 6 (6)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (3) | 4 (5) | 4 (4)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 8 (8) | 6 (6) | 7 (9)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (8) | 15 (17) | 13 (16) | 18 (21)
Sinus pain (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (4) | 2 (2) | 8 (8)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 6 (7)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (5) | 5 (6) | 4 (4)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin urine positive (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reproductive tract disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 5 (5) | 9 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 10 (10) | 7 (8) | 14 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7) | 1 (1) | 8 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 8 (9) | 12 (14) | 18 (19)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 8 (8) | 3 (3) | 5 (5)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hot flashes (Vascular disorders) | 3 (3) | 4 (4) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 6 (8) | 2 (3) | 11 (11)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Thrombosis (Vascular disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Pac --> ddAC) (N=108) | Arm 2 (Pac + Bev --> ddAC + Bev) (N=108) | Arm 3 (Pac + Carboplatin --> ddAC) (N=109) | Arm 4 (Pac + Carboplatin + Bev --> ddAC + Bev) (N=112)
Blood disorder (Blood and lymphatic system disorders) | 75 (196) | 64 (148) | 90 (277) | 92 (255)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 8 (9) | 4 (5) | 11 (11)
Hemoglobin decreased (Blood and lymphatic system disorders) | 9 (20) | 17 (30) | 11 (22) | 12 (31)
Hemolysis (Blood and lymphatic system disorders) | 3 (5) | 1 (1) | 2 (4) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (2) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cardiac pain (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 4 (5) | 8 (10) | 8 (10) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 2 (5) | 3 (5) | 3 (4) | 6 (7)
Stokes-Adams syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 3 (4) | 1 (2) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye syndrome (Eye disorders) | 4 (6) | 3 (3) | 1 (1) | 5 (7)
Eye disorder (Eye disorders) | 4 (6) | 4 (7) | 2 (5) | 1 (2)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flashing vision (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 2 (4) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 14 (23) | 10 (16) | 3 (5) | 13 (24)
Watering eyes (Eye disorders) | 9 (10) | 15 (21) | 8 (9) | 7 (14)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 14 (15) | 5 (8) | 8 (13) | 15 (24)
Anal exam abnormal (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 1 (4)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 1 (2) | 2 (4) | 0 (0) | 1 (1)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 47 (91) | 52 (103) | 47 (88) | 61 (117)
Diarrhea (Gastrointestinal disorders) | 36 (60) | 37 (57) | 33 (52) | 35 (57)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 4 (7) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 28 (43) | 22 (37) | 30 (40) | 30 (51)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 3 (3) | 4 (5) | 3 (3)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 11 (16) | 12 (19) | 14 (16) | 22 (34)
Esophageal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Fistula of small intestine (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (6) | 2 (2) | 2 (2) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 4 (5) | 5 (5) | 1 (1) | 4 (5)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 3 (4) | 4 (4) | 3 (3)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 3 (4) | 7 (9) | 3 (3) | 9 (12)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 22 (37) | 34 (64) | 23 (42) | 30 (52)
Nausea (Gastrointestinal disorders) | 78 (158) | 73 (148) | 74 (173) | 89 (202)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1) | 3 (6) | 5 (5) | 4 (4)
Periodontal disease (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary gland disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 4 (6) | 2 (2) | 1 (1) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Vomiting (Gastrointestinal disorders) | 27 (37) | 28 (37) | 32 (57) | 31 (46)
Chest pain (General disorders) | 4 (6) | 5 (6) | 2 (2) | 2 (2)
Chills (General disorders) | 12 (14) | 8 (9) | 5 (10) | 10 (12)
Edema limbs (General disorders) | 20 (38) | 12 (15) | 12 (19) | 7 (13)
Facial pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 96 (302) | 97 (296) | 97 (293) | 101 (299)
Fever (General disorders) | 13 (13) | 14 (14) | 8 (9) | 10 (13)
Flu-like symptoms (General disorders) | 4 (4) | 2 (4) | 0 (0) | 0 (0)
Gait abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General symptom (General disorders) | 2 (2) | 4 (4) | 0 (0) | 2 (3)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Injection site reaction (General disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Localized edema (General disorders) | 5 (8) | 2 (3) | 2 (2) | 1 (2)
Pain (General disorders) | 17 (32) | 20 (35) | 13 (20) | 18 (22)
Visceral edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic hemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 8 (8) | 11 (12) | 6 (7) | 12 (13)
Immune system disorder (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Bone infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 2 (2)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 4 (4) | 4 (4) | 6 (9) | 4 (8)
Infective myositis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 6 (8) | 7 (8) | 1 (1) | 4 (5)
Otitis externa (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 5 (5) | 3 (3) | 1 (1)
Skin infection (Infections and infestations) | 6 (7) | 11 (14) | 4 (6) | 4 (6)
Soft tissue infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 2 (5) | 4 (6) | 2 (2) | 1 (1)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 5 (5) | 8 (10) | 6 (7) | 8 (9)
Ureteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 9 (11) | 7 (10) | 2 (3) | 10 (11)
Vaginal infection (Infections and infestations) | 2 (2) | 4 (5) | 0 (0) | 1 (1)
Viral hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 3 (4)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 5 (8)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Intraoperative gastrointestinal injury - Teeth (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 7 (12) | 3 (3) | 8 (9)
Alanine aminotransferase increased (Investigations) | 19 (27) | 27 (45) | 22 (43) | 36 (55)
Alkaline phosphatase increased (Investigations) | 13 (24) | 10 (13) | 8 (16) | 17 (34)
Aspartate aminotransferase increased (Investigations) | 20 (36) | 27 (41) | 18 (34) | 29 (44)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 5 (5)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Coagulopathy (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 5 (9) | 2 (5) | 4 (7) | 4 (6)
Electrocardiogram QTc interval prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 5 (5) | 5 (10) | 4 (4) | 8 (12)
Leukocyte count decreased (Investigations) | 23 (45) | 31 (55) | 40 (77) | 39 (81)
Lymphocyte count decreased (Investigations) | 12 (15) | 11 (19) | 8 (11) | 17 (30)
Neutrophil count decreased (Investigations) | 35 (58) | 40 (62) | 85 (173) | 90 (185)
Platelet count decreased (Investigations) | 18 (26) | 19 (29) | 67 (154) | 77 (156)
Serum cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (2)
Weight loss (Investigations) | 10 (12) | 10 (12) | 11 (16) | 18 (23)
Anorexia (Metabolism and nutrition disorders) | 28 (48) | 35 (61) | 33 (58) | 44 (75)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Blood glucose increased (Metabolism and nutrition disorders) | 31 (59) | 28 (49) | 26 (57) | 29 (57)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 6 (8) | 8 (12) | 10 (11) | 11 (13)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 9 (15) | 7 (12) | 6 (7) | 14 (21)
Serum calcium decreased (Metabolism and nutrition disorders) | 13 (18) | 12 (14) | 10 (13) | 9 (12)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (2) | 2 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 2 (2) | 4 (6)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 11 (20) | 2 (2)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 17 (25) | 15 (21) | 28 (57) | 21 (32)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 9 (17) | 12 (20) | 11 (19) | 16 (18)
Serum sodium increased (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 1 (1) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (47) | 23 (39) | 16 (21) | 25 (41)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 11 (15) | 15 (19) | 17 (22)
Bone pain (Musculoskeletal and connective tissue disorders) | 18 (21) | 14 (22) | 8 (10) | 16 (28)
Buttock pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 4 (4) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 0 (0) | 3 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 8 (12) | 2 (7)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (4) | 6 (7) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 36 (58) | 20 (36) | 17 (24) | 25 (48)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (5) | 4 (5) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (22) | 14 (20) | 10 (13) | 9 (10)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0) | 1 (1) | 1 (4)
Arachnoiditis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (3) | 1 (3) | 1 (2)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 3 (4) | 2 (2) | 0 (0) | 3 (3)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 25 (40) | 20 (35) | 22 (31) | 20 (27)
Dysgeusia (Nervous system disorders) | 30 (56) | 22 (43) | 26 (48) | 34 (73)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Headache (Nervous system disorders) | 39 (75) | 45 (77) | 32 (50) | 43 (80)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 3 (6) | 1 (3) | 2 (6) | 2 (2)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 5 (5) | 1 (1) | 4 (5)
Olfactory nerve disorder (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 7 (13) | 10 (16) | 12 (22) | 12 (18)
Peripheral sensory neuropathy (Nervous system disorders) | 80 (221) | 82 (199) | 74 (195) | 83 (178)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (3)
Tremor (Nervous system disorders) | 0 (0) | 3 (6) | 2 (2) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (10)
Anxiety (Psychiatric disorders) | 26 (46) | 18 (34) | 15 (22) | 22 (38)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 20 (35) | 13 (26) | 18 (23) | 17 (28)
Insomnia (Psychiatric disorders) | 34 (72) | 32 (53) | 21 (37) | 30 (57)
Libido decreased (Psychiatric disorders) | 0 (0) | 3 (11) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (1) | 4 (4)
Dysuria (painful urination) (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin urine positive (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 5 (5)
Kidney pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 7 (14) | 1 (1) | 13 (18)
Ureteric hemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 5 (8) | 1 (1) | 3 (3) | 7 (10)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 4 (7) | 1 (1) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Breast pain (Reproductive system and breast disorders) | 10 (15) | 6 (6) | 6 (10) | 5 (8)
Irregular menstruation (Reproductive system and breast disorders) | 2 (3) | 1 (1) | 3 (3) | 6 (10)
Nipple deformity (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reproductive tract disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 2 (3) | 4 (7) | 1 (1) | 2 (3)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 5 (6) | 1 (1) | 3 (3)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 9 (14) | 16 (25) | 8 (11) | 15 (24)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (46) | 31 (61) | 22 (31) | 32 (49)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 38 (63) | 39 (74) | 45 (84) | 48 (93)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 57 (114) | 18 (22) | 58 (97)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 14 (23) | 4 (6) | 9 (10)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 16 (19) | 6 (6) | 10 (16)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 9 (13) | 6 (8) | 8 (11)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 14 (18) | 4 (5) | 13 (25)
Alopecia (Skin and subcutaneous tissue disorders) | 71 (204) | 59 (162) | 55 (136) | 61 (159)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (18) | 18 (26) | 9 (13) | 10 (20)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (6) | 2 (3) | 2 (3)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 6 (7) | 4 (5) | 3 (3) | 3 (5)
Nail disorder (Skin and subcutaneous tissue disorders) | 36 (73) | 38 (74) | 27 (37) | 27 (43)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (22) | 13 (23) | 8 (9) | 12 (16)
Rash acneiform (Skin and subcutaneous tissue disorders) | 11 (21) | 10 (24) | 8 (14) | 9 (10)
Rash desquamating (Skin and subcutaneous tissue disorders) | 26 (45) | 30 (53) | 16 (22) | 19 (29)
Scalp pain (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 6 (10) | 8 (9) | 7 (9) | 11 (14)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (4) | 10 (16) | 5 (7) | 8 (16)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Skin striae (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (4) | 1 (2) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 2 (2)
Sweating (Skin and subcutaneous tissue disorders) | 18 (33) | 4 (7) | 1 (1) | 6 (9)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (5) | 8 (10) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1) | 1 (1) | 2 (3) | 2 (3)
Hot flashes (Vascular disorders) | 32 (82) | 23 (57) | 20 (38) | 19 (40)
Hypertension (Vascular disorders) | 23 (46) | 38 (82) | 11 (16) | 50 (90)
Hypotension (Vascular disorders) | 3 (5) | 3 (4) | 2 (2) | 3 (4)
Lymphedema (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Vascular disorder (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less